CLINICAL TRIAL: NCT01380028
Title: Interest of Oral Corticosteroids in the Treatment of Chronic Subdural Hematomas. Prospective Randomized Multicenter Trial
Brief Title: Interest of Oral Corticosteroids in the Treatment of Chronic Subdural Hematomas
Acronym: hemacort
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: successfull Interim Analysis
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Marseille (Other); Centre Hospitalier Universitaire de Nice (Other); Hospices Civils de Lyon (Other); Centre hospitalier de Perpignan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8545; 2009-015524-28 (EudraCT Number)
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Chronic Intracranial Subdural Hematoma
Keywords: chronic subdural hematomas; corticosteroid; treatment; neurosurgery; recurrence, adjuvant
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence | interventions — Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): The aim of this prospective multicenter randomized, double blind, is to evaluate in patients with chronic subdural hematoma, compared with placebo, the efficacy of postoperative corticosteroid treatment orally for approximately 2 months on the rate of clinical recurrence
  Interventions: Drug: placebo
- oral corticosteroids (Active Comparator): The aim of this prospective multicenter randomized, double blind, is to evaluate in patients with chronic subdural hematoma, compared with placebo, the efficacy of postoperative corticosteroid treatment orally for approximately 2 months on the rate of clinical recurrence
  Interventions: Drug: oral corticosteroids

INTERVENTIONS:
Drug: oral corticosteroids — Active treatment is prednisone establishment within 72 hours after the end of surgery at the dose of 1 mg / kg (rounded to the nearest 10 mg) once daily orally for one week . The daily dose then decreases in increments of 10 mg weekly, by the second week. Once the level of 10 mg / day reached the daily dose by one level lower than 5 mg weekly. Treatment is stopped after this week to 5 mg / day (average 2 months of treatment)
  Other Names: Cortancyl
  Arms: oral corticosteroids
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The chronic subdural hematoma is a common disease in the population over 60 years. For example, in patients over 70 years, it occurs every year 7 new cases per 100,000 people. A chronic subdural hematoma is an accumulation of blood in the intracranial space between brain membrane (dura mater) and the brain. The origin of blood in this area follows a minor brain injury, which causes the rupture of small vessels in the area. During its evolution, the volume of the hematoma increases. After a few weeks, the amount of fluid build-up can compress the brain. That's when clinical symptoms occur: persistent headaches, neurological deficits, seizures, impaired consciousness, cognitive functions (memory loss, impaired intellectual function, or hallucinations, etc.). The compression of the brain may cause impairment of consciousness resulting in more severe cases coma and death. At this stage, a neurosurgical intervention is necessary. Recurrences are numerous (15 to 25% recurrence over six months after neurosurgery). That is why in France, about 20% of medical teams administer a postoperative treatment with corticosteroids to reduce the risk of recurrence. Until now, the potential benefit of this treatment has not yet been confirmed by a clinical study. So the purpose of this research.

DETAILED DESCRIPTION:
The chronic subdural hematoma (HSDC) is a common disease in the population over 60 years. The incidence is 7 / 100000 in patients over 70 years. This condition occurs readily after a minor head injury. Bleeding secondary to cerebral concussion and vascular fragility from a cortico-dural vein. It is favored in most cases by taking anti-platelet or other blood thinners. The hematoma formed and causes a local inflammatory reaction. This reaction tends to partition the collection by the formation of a membrane whose pathological vessels weakened by inflammation, causing bleeding iterative low abundance. A vicious circle is established by a combination of these phenomena and causes a progressive worsening clinical and radiological.Because of the importance of recurrence (15 to 25% at 6 months) and the high rate of mortality at one year (10 to 15%), but also supposed pathophysiological mechanisms (inflammation, formation of membrane self-sustaining blood collection ), a postoperative treatment with corticosteroids was introduced in secondary prevention by some teams (about 20% in France). However, this practice has never been a prospective study on clinical and radiological interest.The aim of this prospective multicenter randomized, double blind, is to evaluate in patients with chronic subdural hematoma, compared with placebo, the efficacy of postoperative corticosteroid treatment orally for approximately 2 months on the rate of clinical recurrence and / or radiological subdural hematoma 6 months after surgery (primary endpoint).The secondary endpoints are the rate of mortality at one year, and the 6 month follow-up of clinical and radiological evolution, neurological status (Markwalder scale), quality of life (health scale perceptual Nottingham), autonomy (Karnofsky scale), the state of consciousness (Glasgow scale), and size of the hematoma on CT scan without injection.340 adult patients of the 2 sexes who received surgical treatment for a chronic subdural hematoma unilateral or bilateral primary diagnosis (hematoma hypodense or isodense with a blade of at least 3 mm thick axial CT scan on brain) will be included in the study on 5 centers (services of Neurosurgery Hospital of Montpellier, Marseille, Nice, Perpignan and Lyon).Patients enrolled will be assigned to one of two treatment groups (active treatment or placebo) by lot. Active treatment is prednisone establishment within 72 hours after the end of surgery at the dose of 1 mg / kg (rounded to the nearest 10 mg) once daily orally for one week . The daily dose then decreases in increments of 10 mg weekly, by the second week. Once the level of 10 mg / day reached the daily dose by one level lower than 5 mg weekly. Treatment is stopped after this week to 5 mg / day .. The placebo was similar in all respects to active treatment and is administered in the same way that the active treatment. Additional treatment will be administered to all patients throughout the duration of the experimental treatment. It is a vitamin and calcium supplementation in preventing the risk of osteoporosis.Medical monitoring of patients will be over a period of six months with visits scheduled in the various departments of Neurosurgery at 1 month, 3 months and 6 months after surgery. Each visit is a consultation with a neurosurgical team physician including a review of clinical research with the recurrence of subdural hematoma and the collection of adverse events. This physician, independent of the investigative team, will also collect scores Markwalder, Nottingham, Karnofsky and Glasgow. Analysis of the CT scan will be centralized. A blood sample will be performed at the visit at 1 month, to establish a biological monitoring in relation to the potential electrolyte disturbances related to steroids.The mortality survey will take place 1 year after surgery by telephone interview between an investigator and the patient or his entourage.The overall duration of the study is about 6 years including 4 years of clinical phase.Given the extensive use of corticosteroids in the treatment of chronic subdural hematomas and absence of solid data on the subject, our research should clarify the role of corticosteroids in secondary prevention and improve the overall management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes operated for chronic subdural hematoma one-sided or bilateral of firstly diagnosis, after consultation in neurosurgery for a symptomatology in touch with this hematic collection.
* At the End of the surgical operation < 72 hours
* Hematoma must be hypodense or isodense. He has to present a value < 50 on the scale of Hounsfield measured in the center of the collection on the initial intellectual scanning, this measure not in front of not to be made on a zone of new bleeding treble or on a membrane (in case of compartmentalized hematoma).

The blade of the hematoma has to measure at least 3 mm in thickness on an axial cutting.

Exclusion Criteria:

* Age < 18 years
* Weight > 104 kg
* Histories of hematoma chronic subdural for which a medical and\or surgical treatment were before realized
* Patient Presenting:

uncontrolled arterial hypertension, current Infection, Diabetes treated by drugs, Ulcer evolutionary gastroduodenal in the course of treatment and dating < 6 months, turned out Osteoporosis symptomatic of cortisone origin, uncontrolled psychotic State by a treatment, except the sultopride, ulcerous Colitis, recent intestinal Anastomose, Renal insufficiency, hepatic Incapacity, Hypercalcemia,Hypercalciuria,calcic Lithiasis, high sensibility at drug'study, Intolerance: galactose, fructose, deficit in lactase, syndrome of malabsorption of glucose or galactose

* Clinical or radiological Characteristics of hematoma suspecting an intra-cranial infection (abscess,..)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-07-22 (Actual); Primary Completion 2014-09-12 (Actual); Study Completion 2014-09-12 (Actual)

PRIMARY OUTCOMES:
the evaluation of efficacy of postoperative corticosteroid treatment in patients group compared with placebo | 6 months after surgery
  The objective of this study is to evaluate in patients with chronic subdural hematoma, compared with placebo, the efficacy of postoperative corticosteroid treatment orally for about two months on the rate of clinical recurrence and / radiological or subdural hematoma 6 months after surgery (primary endpoint).

SECONDARY OUTCOMES:
Evaluation of mortality rate at one year | one year
  Secondary objective is the evaluation of the effectiveness of corticosteroid treatment on the postoperative mortality rate at one year
Evaluation of quality of life at one year | one year
  Secondary objective is the evaluation of the effectiveness of corticosteroid treatment on the quality of life of patients
evaluation of tolerance at one year | one year
  Secondary objective is the evaluation of the tolerance of corticosteroid treatment at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Lonjon Nicolas, MD,PhD, Principal Investigator — CHU de Montpellier
Locations (1):
- Gui de Chauliac Hospital, Montpellier, France